CLINICAL TRIAL: NCT01845311
Title: RESTORE II Trial: Safety & Performance Study of the ReZolve2 Sirolimus-Eluting Bioresorbable Coronary Scaffold
Brief Title: ReZolve2 Clinical Investigation
Acronym: RESTORE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REVA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCT4000
Record Dates: First submitted 2013-03-21; First posted 2013-05-03 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ReZolve2 Treatment Group (Experimental)
  Interventions: Device: ReZolve2 Scaffold

INTERVENTIONS:
Device: ReZolve2 Scaffold

SUMMARY:
The RESTORE II clinical trial is intended to assess safety and performance of the ReZolve2 Bioresorbable Coronary Scaffold in native coronary arteries.

ELIGIBILITY:
Primary Inclusion Criteria:

* Patient has evidence of myocardial ischemia or a positive functional study
* Patient has a normal CK-MB
* Target lesion has a visually estimated stenosis of ≥50% and <100%
* Target lesion is located in a native coronary artery with average reference vessel diameter ≥ 2.75mm and ≤ 3.3mm
* Target lesion length must be ≤ 14mm

Primary Exclusion Criteria:

* Patient has experienced a myocardial infarction (CK-MB or Troponin > 5 X ULN) within 72 hours of the procedure
* Patient has a left ventricular ejection fraction < 30%
* Patient has unprotected lest main coronary disease with ≥50% stenosis
* The target vessel is totally occluded (TIMI Flow 0 or 1)
* Target lesion involves a bifurcation (a lesion with a side branch ≥ 2.0 mm in diameter containing a ≥ 50% stenosis).
* Target lesion is located within a bypass graft
* Target lesion has possible or definite thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 6 Months
Major Adverse Cardiac Events | 12 Months
Late Lumen Loss | 9 Months

SECONDARY OUTCOMES:
QCA derived parameters | 9 Months
  Late Loss, Restenosis Rate, % Diameter Stenosis & Minimum Lumen Diameter
Major Adverse Coronary Events | 24, 36, 48 & 60 Months
  Major Adverse Coronary Events - Combined events consisting of death, myocardial infarction and Target Lesion Revascularization
TLR | 12,24,36,48 & 60 Months
  Target Lesion Revascularization
TVR | 12,24,36,48 & 60 Months
  Target Vessel Revascularization
TVF | 12, 24, 36, 48 & 60 Month
  Target Vessel Failure
Acute Procedural Success | Day 0
  The percentage of patients meeting the Acute Technical Success criteria and the procedure results in a residual stenosis of <50 percent with no immediate (in-hospital) MACE.
Acute Technical Success | Day 0
  The percentage of patients with successful delivery and deployment of the scaffold in the intended lesion without device related complications.
Clinical Procedural Success | 30 Days
  The percentage of patients meeting the Acute Procedural Success criteria with no occurrence of a MACE event through 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; David Muller, MD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (3):
- St Vincent's Hospital, Sydney, Australia
- Instituto Dante Pazzanese de Cariologia, São Paulo, Brazil
- Cardioangiologisches Centrum Bethanien, Frankfurt, Germany